CLINICAL TRIAL: NCT04243577
Title: Development and Validation of Mechanically Compliant Wearable Monitoring Systems for Swallowing Function and Disorders
Brief Title: Wearable Monitoring Systems for Swallowing Function and Disorders
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Georgia A. Malandraki, Associate Professor, Department of Speech, Language and Hearing Sciences, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1807020788; 1R21EB026099-01A1 (NIH)
Record Dates: First submitted 2019-08-26; First posted 2020-01-28 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: Deglutition Disorders
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Experiments will follow a within-subject randomized cross-over design. The purpose is to develop devices that are optimized for their use. To achieve this goal, for each new iteration of the devices, at least ten new participants will be tested using the current prototypes and the commercially available counterpart sensors in counterbalanced order. Results will be analyzed and discussed in regards to design improvements before the next iteration of development. The plan to recruit a large number of total subjects allows for several pre-clinical experiments to be conducted until the final versions of both devices are optimized.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Group A: Conventional Sensors First, Then Experimental (Tele-EaT) Sensors (Other): Group A participants will complete the experimental protocol (swallow trials) with the conventional (commercially available) electrodes/sensors first. After a break of 10 minutes, they then will repeat the exact same experimental protocol (exact same swallow trials) with the experimental sensors (i.e., a wearable surface EMG sensors patch we are developing).
  Interventions: Device: Tele-EaT Sensors; Device: Conventional Sensors
- Group B: Experimental (Tele-EaT) Sensors First, Then Conventional Sensors (Other): Group B participants will complete the experimental protocol (swallow trials) with the experimental sensors (i.e., a wearable surface EMG sensors patch we are developing) first. After a break of 10 minutes, they then will repeat the exact same experimental protocol (exact same swallow trials) with the conventional (commercially available) electrodes/sensors.
  Interventions: Device: Tele-EaT Sensors; Device: Conventional Sensors

INTERVENTIONS:
Device: Tele-EaT Sensors — Two iterations of a wearable surface EMG (sEMG) sensors patch we developed will be tested against commercially available wired devices. The first iteration of the wearable sensor patch is an ultrathin patch with a honeycomb-inspired design that included sEMG and strain sensors in order to capture muscle activity and thyroid movement signals from the submental area during swallows and swallow maneuvers/exercises. The second iteration is a more durable slightly thicker flexible, non-stretchable, and double-sided thin sEMG patch. Participants will perform standardized swallow tasks while wearing the device.
Device: Conventional Sensors — Conventional sensors will include snap-on wired electrodes as the control condition. The same set of standardized swallow tasks will be completed with the conventional and commercially available devices as well.

SUMMARY:
Wearable tele-rehabilitation technology allows for the efficient provision of rehabilitation services from a distance, facilitating tele-management of many disorders. The proposed research will develop and validate a set of mechanically compliant, easy-to-use, and inexpensive wearable tele-monitoring systems, for future use in the rehabilitation of swallowing disorders (dysphagia). The hypothesis is that the newly developed wearable sensors will have equal or better performance than traditional wired sensors used today in clinical practice. Factors related to signal quality and patient reported outcomes (e.g., satisfaction/comfort level, adverse effects etc.) will be examined.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for healthy adults:

* Age 18-30 OR 50-90 years of age
* No history of dysphagia
* No history of a neurological disorder
* A score in the normal/mild range on the Montreal Cognitive Assessment (MoCA):
* A score of <3 on the Eating Assessment Tool-10 (EAT-10, a self-report screening for dysphagia).

Inclusion criteria for patients with dysphagia:

* Age 18-90 years of age
* Diagnoses of dysphagia as a result of a neurological disorder (e.g., stroke, Parkinson's disease).
* A score in the normal/mild range on the Montreal Cognitive Assessment (MoCA).
* A score of ≥3 on the Eating Assessment Tool-10 (EAT-10, a self-report screening for dysphagia).

Exclusion Criteria:

• Significant cognitive impairment (a score in the moderate-severe range on MoCA):

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georgia A. Malandraki, PhD, Principal Investigator — Professor; Chi Hwan Lee, PhD, Principal Investigator — Associate Professor
Locations (1):
- Purdue University I-EaT Lab, West Lafayette, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two iterations of the sensors were tested against commercial sensors. For iteration 1, 51 healthy older adults were screened for eligibility between September and November 2018. For iteration 2, 38 healthy older adults were screened for eligibility between October 2021 and March 2023. All was completed at a university research lab and clinic in West Lafayette, Indiana.
Pre-assignment Details: For iteration 1, 40 of the 51 participants were randomized into one of 2 groups for testing 1. Of those not randomized, 7 did not meet inclusion criteria, 1 declined to participate, and 1 did not participate due to other reasons (scheduling conflicts or technical issues).
  For iteration 2, 30 of the 38 participants were randomized into one of 2 groups for testing 2. Of those not randomized, 7 did not meet inclusion criteria, and 1 did not participate due to other reasons (technical issues).
Groups:
- Group A1: Conventional Sensors First, Then Experimental (Tele-EaT) Sensors - Iteration 1: Group A1 participants completed the experimental protocol (swallow trials) with the conventional (commercially available) electrodes/sensors first. After a break of 10 minutes, they then repeated the exact same experimental protocol (exact same swallow trials) with the first iteration of the experimental sensors (i.e., a wearable surface EMG sensors patch we are developing).
  Tele-EaT Sensors - Iteration 1: A first iteration of a wearable surface EMG (sEMG) sensors patch we developed was tested against commercially available wired devices. The first iteration of the wearable sensor patch is an ultrathin patch with a honeycomb-inspired design that included sEMG and strain sensors in order to capture muscle activity and thyroid movement signals from the submental area during swallows and swallow maneuvers/exercises. Participants performed standardized swallow tasks while wearing the first iteration device.
  Conventional Sensors: Conventional sensors included snap-on wired electrodes as the control condition. The same set of standardized swallow tasks was completed with the conventional and commercially available devices as well.
- Group B1: Experimental (Tele-EaT) Sensors - Iteration 1 First, Then Conventional Sensors: Group B1 participants completed the experimental protocol (swallow trials) with the first iteration of the experimental sensors (i.e., a wearable surface EMG sensors patch we are developing) first. After a break of 10 minutes, they then repeated the exact same experimental protocol (exact same swallow trials) with the conventional (commercially available) electrodes/sensors.
  Tele-EaT Sensors -Iteration 1: The first iteration of a wearable surface EMG (sEMG) sensors patch we developed was tested against commercially available wired devices. The first iteration of the wearable sensor patch is an ultrathin patch with a honeycomb-inspired design that included sEMG and strain sensors in order to capture muscle activity and thyroid movement signals from the submental area during swallows and swallow maneuvers/exercises. Participants performed standardized swallow tasks while wearing the device.
  Conventional Sensors: Conventional sensors included snap-on wired electrodes as the control condition. The same set of standardized swallow tasks was completed with the conventional and commercially available devices as well.
- Group A2: Conventional Sensors First, Then Experimental (Tele-EaT) Sensors - Iteration 2: Group A2 participants completed the experimental protocol (swallow trials) with the conventional (commercially available) electrodes/sensors first. After a break of 10 minutes, they then repeated the exact same experimental protocol (exact same swallow trials) with the second iteration of the experimental sensors (i.e., a wearable surface EMG sensors patch we are developing).
  Tele-EaT Sensors - Iteration 2: A second improved iteration of a wearable surface EMG (sEMG) sensors patch we developed was tested against commercially available wired devices. The second iteration of the wearable sensor patch is a more durable slightly thicker flexible, non-stretchable, and double-sided thin sEMG patch. Participants performed standardized swallow tasks while wearing the second iteration device.
  Conventional Sensors: Conventional sensors included snap-on wired electrodes as the control condition. The same set of standardized swallow tasks was completed with the conventional and commercially available devices as well.
- Group B2: Experimental (Tele-EaT) Sensors - Iteration 2 First, Then Conventional Sensors: Group B2 participants completed the experimental protocol (swallow trials) with the second iteration of the experimental sensors (i.e., a wearable surface EMG sensors patch we are developing) first. After a break of 10 minutes, they then repeated the exact same experimental protocol (exact same swallow trials) with the conventional (commercially available) electrodes/sensors.
  Tele-EaT Sensors - Iteration 2: The second improved iteration of a wearable surface EMG (sEMG) sensors patch we developed was tested against commercially available wired devices. The second iteration of the wearable sensor patch is a more durable slightly thicker flexible, non-stretchable, and double-sided thin sEMG patch. Participants performed standardized swallow tasks while wearing the device.
  Conventional Sensors: Conventional sensors included snap-on wired electrodes as the control condition. The same set of standardized swallow tasks was completed with the conventional and commercially available devices as well.
Period: First Intervention (1 Hour)
Arm/Group | Group A1: Conventional Sensors First, Then Experimental (Tele-EaT) Sensors - Iteration 1 | Group B1: Experimental (Tele-EaT) Sensors - Iteration 1 First, Then Conventional Sensors | Group A2: Conventional Sensors First, Then Experimental (Tele-EaT) Sensors - Iteration 2 | Group B2: Experimental (Tele-EaT) Sensors - Iteration 2 First, Then Conventional Sensors
Started | 20 | 20 | 15 | 15
Completed | 20 | 20 | 15 | 15
Not Completed | 0 | 0 | 0 | 0
Period: Washout (10 Minutes)
Arm/Group | Group A1: Conventional Sensors First, Then Experimental (Tele-EaT) Sensors - Iteration 1 | Group B1: Experimental (Tele-EaT) Sensors - Iteration 1 First, Then Conventional Sensors | Group A2: Conventional Sensors First, Then Experimental (Tele-EaT) Sensors - Iteration 2 | Group B2: Experimental (Tele-EaT) Sensors - Iteration 2 First, Then Conventional Sensors
Started | 20 | 20 | 15 | 15
Completed | 20 | 20 | 15 | 15
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention (1 Hour)
Arm/Group | Group A1: Conventional Sensors First, Then Experimental (Tele-EaT) Sensors - Iteration 1 | Group B1: Experimental (Tele-EaT) Sensors - Iteration 1 First, Then Conventional Sensors | Group A2: Conventional Sensors First, Then Experimental (Tele-EaT) Sensors - Iteration 2 | Group B2: Experimental (Tele-EaT) Sensors - Iteration 2 First, Then Conventional Sensors
Started | 20 | 20 | 15 | 15
Completed | 20 | 20 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A1: Conventional Sensors First, Then Experimental (Tele-EaT) Sensors - Iteration 1 | Group B1: Experimental (Tele-EaT) Sensors - Iteration 1 First, Then Conventional Sensors | Group A2: Conventional Sensors First, Then Experimental (Tele-EaT) Sensors - Iteration 2 | Group B2: Experimental (Tele-EaT) Sensors - Iteration 2 First, Then Conventional Sensors | Total
Number analyzed (Participants) | 20 | 20 | 15 | 15 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.5 (8.8) | 68.3 (6.7) | 63.6 (10) | 65.7 (8.4) | 66.3 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 7 | 6 | 29
  Male | 15 | 9 | 8 | 9 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 15 | 13 | 68
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 19 | 20 | 15 | 12 | 66
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 15 | 15 | 70

OUTCOME MEASURES:

1. Primary Outcome: Normalized Task-related sEMG Amplitude (Signal Quality Parameter)
Description: Normalized sEMG amplitude values during standardized swallow tasks and maneuvers will be recorded and compared between the two sEMG devices. Normalized amplitude is used as a signal quality parameter and is not a health related outcome.
Time Frame: Post each experiment (i.e., 1 hour after the sensors have been placed)
Population: Reminder: The first iteration testing of the Tele-EaT sensors was tested against commercial/conventional sensors in 40 participants. The second iteration testing was tested in an additional 30 participants.
Measure: Mean (Standard Deviation); unit: percentage of maximum amplitude
Groups:
- Conventional Sensors - Iteration Testing 1: Outcomes measured while using the conventional sensors during iteration testing 1 .
- Tele-EaT Sensors - Iteration Testing 1: Outcomes measured while using the first version of the experimental (Tele-EaT) sensors during iteration testing 1.
- Conventional Sensors - Iteration Testing 2: Outcomes measured while using the conventional sensors during iteration testing 2.
- Tele-EaT Sensors - Iteration Testing 2: Outcomes measured while using the second version of the experimental (Tele-EaT) sensors during iteration testing 2.
Arm/Group | Conventional Sensors - Iteration Testing 1 | Tele-EaT Sensors - Iteration Testing 1 | Conventional Sensors - Iteration Testing 2 | Tele-EaT Sensors - Iteration Testing 2
Number analyzed (Participants) | 40 | 40 | 30 | 30
percentage of maximum amplitude | 12.5 (7) | 11.7 (7.3) | 17.3 (8) | 13.8 (6.2)
Statistical Analysis 1: Comparison: Conventional Sensors - Iteration Testing 1 vs Tele-EaT Sensors - Iteration Testing 1; For Iteration 1 testing, we hypothesized that normalized amplitude during swallow trials obtained using the conventional sensors and the experimental sensors will be equivalent. Alpha level was set to .025 to correct for multiple comparisons; Test type: Equivalence — Margins for this test were calculated as plus or minus half a standard deviation using preliminary data acquired with the conventional electrodes, which were considered as the current gold standard and were ± 3.1; p < 0.025, t-test, 2 sided — Alpha level based on Bonferroni correction was set to .025 to correct for multiple comparisons
Statistical Analysis 2: Comparison: Conventional Sensors - Iteration Testing 2 vs Tele-EaT Sensors - Iteration Testing 2; For Iteration 2 testing again, we hypothesized that normalized amplitude during swallow trials obtained using the conventional sensors and the experimental sensors will be equivalent. Alpha level was set to .025 to correct for multiple comparisons; Test type: Equivalence — Margins for this test were based on the absolute value of the effect size (Cohen's d) being smaller than 0.5; p < 0.025, Bootstrapping CIs — Alpha level based on Bonferroni correction was set to .025 to correct for multiple comparisons; In this 2nd iteration testing, we are accounting for variance uncertainty, and thus bootstrapping a Confidence Interval for Cohen's d

2. Primary Outcome: Signal to Noise Ratio (Signal Quality Parameter)
Description: Signal to Noise ratio will be calculated and compared between sensor types tested. Signal to noise ration is a signal quality parameter and not a health related outcome.
Time Frame: Post each experiment (i.e., 1 hour after the sensors have been placed)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Signal to noise ratio
Arm/Group | Conventional Sensors - Iteration Testing 1 | Tele-EaT Sensors - Iteration Testing 1 | Conventional Sensors - Iteration Testing 2 | Tele-EaT Sensors - Iteration Testing 2
Number analyzed (Participants) | 40 | 40 | 30 | 30
Signal to noise ratio | 19.5 (5.2) | 20.4 (5) | 25.1 (5.5) | 26.7 (3.9)
Statistical Analysis 1: Comparison: Conventional Sensors - Iteration Testing 1 vs Tele-EaT Sensors - Iteration Testing 1; For Iteration 1 testing, we hypothesized that Signal to Noise Ratio (SNR) obtained using the experimental sensors will not be inferior to the Signal to Noise Ratio (SNR) obtained using the conventional sensors. Alpha level was set to .025 to correct for multiple comparisons; Test type: Non-Inferiority — Margin for this test was calculated as minus half a standard deviation using preliminary data acquired with the conventional electrodes, which were considered as the current gold standard and was -.99; p < 0.025, t-test, 1 sided — Alpha level based on Bonferroni correction was set to .025 to correct for multiple comparisons
Statistical Analysis 2: Comparison: Conventional Sensors - Iteration Testing 2 vs Tele-EaT Sensors - Iteration Testing 2; For Iteration 2 testing, we again hypothesized that Signal to Noise Ratio (SNR) obtained using the newer version of the experimental sensors will not be inferior to the Signal to Noise Ratio (SNR) obtained using the conventional sensors. Alpha level was set to .025 to correct for multiple comparisons; Test type: Non-Inferiority — Margin for this test was based on the effect size (Cohen's d) being larger than -0.5; p < 0.025, Bootstrapping CIs — Alpha level based on Bonferroni correction was set to .025 to correct for multiple comparisons; In this 2nd iteration testing, we are accounting for variance uncertainty, and thus bootstrapping a one-sided confidence bound for Cohen's d

3. Secondary Outcome: Ease of Use/Comfort
Description: Ease-of-use/comfort will be examined using a survey also devised by the investigators (using a positive centered 5-point Likert scale) with questions about ease-of-use/comfort after each experiment with each device. This survey includes statements related to the participants' ease-of-use/comfort during the experimental protocol (e.g., I was comfortable while the experimenter placed the sensors on my skin). The answers will be rated on a 10-point scale (i.e., 1 = extremely uncomfortable, 10 = extremely comfortable). Higher values indicate better or higher satisfaction/comfort scores. Total scores will be compared across conditions/devices tested.
  For the first iteration testing, the scale used for this outcome measure included 5 survey questions rated on a 10-point scale (total possible: 50; range 0-50). For the second iteration testing, we added one more question, hence the scale included 6 survey questions (total possible: 60; range: 0-60).
Time Frame: Post each experiment (i.e., 1 hour after the sensors have been placed)
Population: The first iteration test of the Tele-EaT sensors against commercial/conventional sensors included 40 participants. The second iteration testing was tested in an additional 30 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Conventional Sensors - Iteration Testing 1 | Tele-EaT Sensors - Iteration Testing 1 | Conventional Sensors - Iteration Testing 2 | Tele-EaT Sensors - Iteration Testing 2
Number analyzed (Participants) | 40 | 40 | 30 | 30
score on a scale | 48.06 (3.6) | 48.62 (3.2) | 54 (8.3) | 57 (4.2)
Statistical Analysis 1: Comparison: Conventional Sensors - Iteration Testing 1 vs Tele-EaT Sensors - Iteration Testing 1; For Iteration 1 testing, we hypothesized that ease of use/comfort expressed after using the experimental patch will be higher than the one reported using the conventional electrodes. Alpha level was set to .05; Test type: Superiority; p < 0.05, t-test, 1 sided; Paired t-test
Statistical Analysis 2: Comparison: Conventional Sensors - Iteration Testing 2 vs Tele-EaT Sensors - Iteration Testing 2; For Iteration 2 testing, again we hypothesized that ease of use/comfort expressed after using the experimental patch will be higher than the one reported using the conventional electrodes. Alpha level was set to .05; Test type: Superiority; p < 0.05, t-test, 1 sided; Paired t-test

4. Secondary Outcome: Adverse Effects and Safety
Description: Safety will be examined by documenting the incidence of skin irritations and pain in the subjects. A visual inspection form including a binary scale (YES/NO) has been devised by the investigators (no formal name) and will be used by a rater who will thoroughly inspect the participants' submandibular skin before and after each experiment. For any irritation or change in appearance YES will be selected and the type of irritation will be descriptively recorded (e.g., red skin). Pain is also rated in the same way through a question to the participants. This form will be completed by a rater who is not part of the data collection process and who is blinded to sensors type to avoid any bias.The number of YESs will be used to calculate the incidence of these adverse effects in the sample.
Time Frame: Pre and Post each experiment (i.e., right before the placement of sensors on the subject and 1 hour after the sensors have been placed and 5 minutes after their removal)
Population: Reminder: The first iteration testing of the Tele-EaT sensors was tested against commercial/conventional sensors in 40 participants. The second iteration testing was tested in an additional 30 participants. For this outcome measure, cumulative data across both time points are presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional Sensors - Iteration Testing 1 | Tele-EaT Sensors - Iteration Testing 1 | Conventional Sensors - Iteration Testing 2 | Tele-EaT Sensors - Iteration Testing 2
Number analyzed (Participants) | 40 | 40 | 30 | 30
Participants | 8 | 1 | 12 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data were collected immediately after removal of each sensors type (post each experiment) and 5 minutes later as well.
Description: We collected potential adverse data on two relevant factors: skin irritation and pain.
  For skin irritation, a YES/NO binary visual inspection/observation form was completed for each of three items: redness, skin irritation, itchiness.
  For pain, a YES/NO binary observation form was completed. If the answer was yes at any point, the participants were asked to rate the pain level as well on a scale from 0-10.
Arm/Group | Conventional Sensors - Iteration Testing 1 | Tele-EaT Sensors - Iteration Testing 1 | Conventional Sensors - Iteration Testing 2 | Tele-EaT Sensors - Iteration Testing 2
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 8/40 | 1/40 | 12/30 | 4/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Sensors - Iteration Testing 1 (N=40) | Tele-EaT Sensors - Iteration Testing 1 (N=40) | Conventional Sensors - Iteration Testing 2 (N=30) | Tele-EaT Sensors - Iteration Testing 2 (N=30)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) — For skin irritation, a YES/NO binary visual inspection/observation form was completed. If any skin irritation (other than redness) was reported by the participant either immediately after removal of sensors or 5 minutes later, this was recorded.
Skin redness (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 6 (6) | 2 (2) — For skin redness, a YES/NO binary visual inspection/observation form was completed. If any skin redness was visually inspected either immediately after removal of sensors or 5 minutes later, this was recorded.
Itchiness (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) — For itchiness, a YES/NO binary visual inspection/observation form was completed. If any itchiness was reported by the participant either immediately after removal of sensors or 5 minutes later, this was recorded.
Pain (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) — For pain, a YES/NO binary observation form was completed. If the answer was yes at any point, the participants were asked to rate the pain level as well on a scale from 0-10.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT04243577/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT04243577/ICF_001.pdf